CLINICAL TRIAL: NCT01638091
Title: Practice-Based Learning to Predict Polyp Histology at Colonoscopy: A Demonstration Project in Community Practice
Brief Title: Practice-Based Learning to Predict Polyp Histology at Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HSR-10-1167; IRB-20373 (Other: Stanford University IRB)
Record Dates: First submitted 2012-07-06; First posted 2012-07-11 (Estimated); Last update posted 2012-07-11 (Estimated); Status verified 2012-07

CONDITIONS: Colonic Polyps; Adenomatous Polyps
Keywords: Narrow band imaging; Screening colonoscopy; Histology
MeSH Terms: conditions — Colonic Polyps; Adenomatous Polyps

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All participating endoscopists (Experimental): All endoscopists will undergo ex vivo training and will participate in in vivo practice-based learning.
  Interventions: Behavioral: Ex vivo module; Behavioral: In vivo practice-base learning phase

INTERVENTIONS:
Behavioral: Ex vivo module — Pre-test, ex vivo computerized training module, post-test
Behavioral: In vivo practice-base learning phase — Prediction of polyp histology in real time, comparison to pathology reports, and review of cumulative individual performance.

SUMMARY:
Most colorectal cancers arise from polyps. Most polyps removed at colonoscopy are small. New technologies such as narrowband imaging (NBI) offer the possibility of in differentiation between precancerous and unimportant small polyps. Use of these technologies could decrease the costs and potentially the risks of screening and surveillance colonoscopy.

Multiple studies have demonstrated the ability of experienced endoscopists to achieve high accuracy in differentiating polyp types using NBI.

The investigators hypothesize that community-based endoscopists can learn to identify polyp type at colonoscopy with the aid of NBI through the use of an introductory didactic program, followed by practice based-learning, and that their experience can serve as guidelines for wider dissemination.

The purpose of this study is to test an educational program combining a didactic program followed by practice-based learning that is designed to allow community-based endoscopists to become proficient at the use of NBI in the colon. This study will not affect the care of patients in any way. The research subjects will be the endoscopists, who will perform colonoscopy and polyp removal in the usual clinical fashion, with the addition of attempting to predict polyp type before resection.

DETAILED DESCRIPTION:
A) Study Purpose and Rationale Most polyps removed at colonoscopy are small. The natural history of these polyps is not understood completely, but the risk of subsequent cancer in persons with small rectosigmoid adenomas may not be higher than in persons without rectosigmoid adenomas [1]. With improvements in colonoscopic imaging, experienced endoscopists can detect polyps in a large fraction of patients. Removal of all small polyps followed by formal histopathological examination increases the costs associated with colorectal cancer screening, and may increase the risk of complications, depending on the technique that is used for polypectomy.

New technologies such as narrowband imaging (NBI) offer the possibility of in vivo differentiation between adenomatous and hyperplastic polyps. Policies to leave in place small polyps that appear to be hyperplastic, or to remove and discard small polyps after in vivo histologic categorization without formal histopathology review could significantly decrease the costs and potentially the risks of screening and surveillance colonoscopy.

Multiple studies have demonstrated the ability of experienced endoscopists to achieve high accuracy in differentiating adenomatous from hyperplastic polyps using NBI [2, 3, 4, 5]. The level of confidence associated with in vivo histologic categorization of a particular polyp is a valuable adjunct measure in determining subsequent clinical management. Dissemination to the community setting of policies that promote in vivo histologic categorization is likely to require practice-based learning.

B) Hypotheses The investigators hypothesize that community-based endoscopists can learn to identify polyp histology at colonoscopy with the aid of NBI through the use of an introductory didactic program, followed by practice based-learning, and that representative learning curves can be generated that can serve as guidelines for wider dissemination.

C) Purpose The purpose of this study is to test an educational program combining a didactic program followed by practice-based learning that is designed to allow community-based endoscopists to become proficient at in vivo histologic characterization of small polyps with the aid of NBI. This study will not require any changes in endoscopists' decisions regarding the indications and methods for polypectomy.

This study will not address directly whether polyps predicted to be hyperplastic or even diminutive adenomas should be left in place, or discarded and not submitted for formal histopathological review.

D) Specific Aims This study has two primary and two secondary aims

1. One primary aim is to assess the proficiency of community-based endoscopists at ex vivo histologic characterization of polyps using NBI based on photographs before and after a didactic program designed to familiarize them with in vivo histologic characterization.
2. The central primary aim is to assess whether the currently designed program is effective at training endoscopists to classify adenomatous vs. hyperplastic polyps in practice with at least 90% accuracy.
3. A secondary aim is to characterize endoscopists' individual and group average learning curves for in vivo histologic characterization using NBI during practice-based learning, with attention to level of confidence, accuracy, sensitivity, specificity and positive and negative predictive values.
4. Another secondary aim is to determine whether surveillance recommendations that would be made based on in vivo histologic characterization using NBI are comparable to those based on formal histopathological assessment.

E) Timeline for assessments:

Endoscopists' accuracy will be determined at three pre-specified points: after assessment of 50, 70 and 90 independent diminutive polyps (defined as <=5mm polyps, one per study colonoscopy, with random selection in cases of >1 diminutive polyp per study colonoscopy). We estimate that in order to assess 90 independent diminutive polyps, endoscopists will need to participate for 6-12 months.

ELIGIBILITY:
Inclusion Criteria:

* Community-based endoscopist who performs screening colonoscopy

Exclusion Criteria:

* Inability or lack of willingness to provide informed consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-03; Primary Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Proportion of participants achieving 90% accuracy | 6-12 months depending on when an endoscopist has assessed 50, 70 and 90 independent diminutive polyps
  Success for a participant was defined as achieving ≥90% accuracy in optical diagnosis of diminutive polyps. This was based on the last 30 consecutive independent diminutive polyps per participant at one of three pre-specified points (at polyp #50, 70 or 90).

SECONDARY OUTCOMES:
Learning curves | 6-12 months depending on when an endoscopist has assessed 50, 70 and 90 independent diminutive polyps
  Leraning curves as a function of polyp batch, for sensitivity, specificity, positive and negative predictive values, and accuracy
Surveillance recommendations | 6-12 months depending on when an endoscopist has assessed 50, 70 and 90 independent diminutive polyps
  Agreement between NBI-aided surveillance recommendations vs. those based on pathology examination of all polyps

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Stanford University, Stanford, California
  - Huron Gastroenterology, Ann Arbor, Michigan

REFERENCES:
- [Derived] Ladabaum U, Fioritto A, Mitani A, Desai M, Kim JP, Rex DK, Imperiale T, Gunaratnam N. Real-time optical biopsy of colon polyps with narrow band imaging in community practice does not yet meet key thresholds for clinical decisions. Gastroenterology. 2013 Jan;144(1):81-91. doi: 10.1053/j.gastro.2012.09.054. Epub 2012 Oct 3. PMID 23041328